CLINICAL TRIAL: NCT07109843
Title: Effect of Boswellia Serrata on Pain Intensity, Central and Peripheral Sensitization, and Pain Modulation in Healthy Volunteers - a Randomized, Double-blind, Placebo-controlled, Cross-over Pilot Trial
Brief Title: Effect of Boswellia Serrata on Pain Intensity, Central and Peripheral Sensitization, and Pain Modulation in Healthy Volunteers
Acronym: BSPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BS2025PP; Medical University of Graz (Other: Medical University of Graz)
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Central Sensitisation; Peripheral Sensitization; Neuroinflammatory Response
MeSH Terms: conditions — Chronic Pain | interventions — Frankincense

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Boswellia Serrata) (Experimental): One capsule 600mg per day for 28 days
  Interventions: Dietary Supplement: Boswellia serrata extract; Other: Placebo
- Placebo (Placebo Comparator): 1 capsule placebo per day for 28 days
  Interventions: Dietary Supplement: Boswellia serrata extract; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Boswellia serrata extract — Boswellia Serrata 1x day (600mg)
  Other Names: Boswellia
Other: Placebo — Placebo 1x/day

SUMMARY:
This planned study is based on a randomized, placebo-controlled cross-over design.

Boswellic acids, the triterpenes found in the gum resins of Boswellia serrata (family: Burseraceae), are traditionally used in the Indian Ayurvedic medicine system as antioxidants and anti-inflammatory agents for treating conditions such as rheumatoid arthritis, chronic bronchitis, asthma, and chronic inflammatory bowel diseases (ulcerative colitis and Crohn's disease). The β-configured pentacyclic triterpenic acids in B. serrata include 3-acetyl-11-keto-β-boswellic acid (AKBBA), 11-keto-β-boswellic acid (KBBA), β-boswellic acid (BBA), and 3-acetyl-β-boswellic acid (ABBA). These compounds, which constitute approximately 14% of the lipophilic fractions of the B. serrata extract, are the major active components. Boswellia serrata is marketed as a food supplement in accordance with EU Directive 2002/46/EC. Several clinical studies have examined the efficacy of B. serrata in chronic pain conditions.

The data suggest a clinical analgesic efficacy, without, however, allowing conclusions about the underlying mechanisms. These have not yet been investigated in a human experimental pain model. The aim of the study is to investigate the influence of Boswellia serrata in peripheral and central sensitization, as well as descending inhibitory pathways by Quantitative Sensory Testing (QST). These findings are of great relevance for a better understanding of clinical efficacy.

The 'Capsaicin Pain Model' is a validated method for inducing short-term peripheral and central sensitization. As a non-invasive human pain model, it is therefore well suited for investigating the analgesic and anti-hyperalgesic effects of drugs.

Furthermore, the influence of Boswellia serrata on mood (depression, anxiety), sleep quality and psychological well-being will be investigated by using the psychological questionnaires Becks-Depression-Inventory, Becks-Anxiety-Inventory, Pittsburgh Sleep Quality Index and World Health Organization Well-Being Index (BDI-II, BAI, PSQI and WHO5) as secondary target variables.

DETAILED DESCRIPTION:
"Boswellic acids, the triterpenes found in the gum resins of Boswellia serrata (family: Burseraceae), are traditionally used in the Indian Ayurvedic medicine system as antioxidants and anti-inflammatory agents for treating conditions such as rheumatoid arthritis, chronic bronchitis, asthma, and chronic inflammatory bowel diseases (ulcerative colitis and Crohn's disease).

The β-configured pentacyclic triterpenic acids in B. serrata include 3-acetyl-11-keto-β-boswellic acid (AKBBA), 11-keto-β-boswellic acid (KBBA), β-boswellic acid (BBA), and 3-acetyl-β-boswellic acid (ABBA). These compounds, which make up about 14% of the lipophilic fractions of B. serrata extract, are the major active components. Various pharmacological studies suggest that the β-configured derivatives of boswellic acids from BSE exhibit significantly better efficacy than their corresponding α-isomers. Additionally, the anti-inflammatory effects of BSE are well-documented in animal models, particularly in the inhibition of carrageenan-induced paw edema.

The data suggest a clinical analgesic efficacy, without, however, allowing conclusions about the underlying mechanisms. These have not yet been investigated in a human experimental pain model. The aim of the study is to investigate the influence of B. serratain peripheral and central sensitization, as well as descending inhibitory pathways by Quantitative Sensory Testing (QST). These findings are of great relevance for a better understanding of clinical efficacy.

An effect on peripheral sensitization speaks in favor of use in acute somatic pain. However, if the effect can be explained by central mechanisms, its use would be recommended in chronic or neuropathic pain. For this purpose, "Capsaicin Pain model" is a validated method for achieving short-term peripheral and central sensitization. As a non-invasive human pain model, it is therefore well suited for investigating the analgesic and anti-hyperalgesic effects of drugs.

Furthermore, the influence of B. serrata on mood (depression, anxiety), sleep quality and psychological well-being will be investigated by using the psychological questionnaires Becks-Depression-Inventory, Becks-Anxiety-Inventory, Pittsburgh Sleep Quality Index and World Health Organization Well-Being Index (BDI-II, BAI, PSQI and WHO5) as secondary target variables.

The following questions were be answered in this study:

Can the administration of Boswellia serrata reduce spontaneous pain following repetitive phasic heat application? Does the intake of Boswellia serrata modulate central sensitization? Does the intake of Boswellia serrata influence peripheral sensitization? Can the descending inhibitory pathways be modulated through the administration of Boswellia serrata? Is a reduction in depression scores achievable through Boswellia serrataadministration? Can anxiety scores be reduced by the administration of Boswellia serrata? Is sleep quality improved with the intake of Boswellia serrata?

The following methods were used to answer these questions:

Spontaneous pain was determined using the numeric rating scale (NRS). Central sensitization was evaluated by pain sensitivity to mechanical stimuli, i.e. pinprick hyperalgesia or allodynia.

An effect on peripheral sensitization was investigated by measuring the heat detection threshold and heat pain threshold.

The body's own pain inhibition was evaluated by means of a "conditioned pain modulation" test.

The influence on mood (depression, anxiety), sleep quality and psychological well-being were evaluated using psychological questionnaires (BDI-II, BAI, PSQI and WHO5).

The intake of Boswellia serrata 2 x 300 mg over 28 days does not change the spontaneous pain after repetitive phasic heat application compared to placebo intake.

Alternative hypothesis:

The intake of Boswellia serrata 2x 300 mg over 28 days changes the spontaneous pain after repetitive phasic heat application compared to placebo intake.

Secondary hypotheses:

There is a significant difference in the size of the mechanical allodynia distance and the flare area after repetitive phasic heat application when taking Boswellia serrata compared to placebo.

There is a change in pinprick hyperalgesia with Boswellia serrata compared to placebo after repetitive phasic heat application.

The intake of Boswellia serrata leads to a change in the heat perception and pain threshold compared to placebo intake after repetitive phasic heat application.

The intake of Boswellia serrata leads to a change in "conditioned pain modulation" compared to placebo intake.

Study design:

This study is based on a pilot, randomized, double-blind, placebo-controlled, cross-over design.

After recruitment, information and inclusion of the study participants, the first baseline measurement consisting of the sensory parameters is carried out. The test subjects are randomized into two groups. They take either the test substance (verum; 600 mg Boswellia serrata daily) or the placebo for 28 days. Both the participants and the study staff responsible for collecting the measurement parameters are blinded to the order in which the tablets are taken.

After recruitment, information and inclusion of the subjects in the study, the first baseline measurement is performed. After 28 days, during which either the verum or study substance is taken, the influence on the "conditioned pain modulation" is measured. The "Capsaicin pain model" according to the published procedures follows. In this trial, the heat/capsaicin model will be used without intradermal injection to further minimize the risk of skin injury, while still inducing painful stimuli and long-lasting cutaneous hyperalgesia. By using a patch, we avoid the extreme pain intensity associated with intradermal capsaicin injection.

Local administration of capsaicin to human skin rapidly leads to a local neurogenic inflammation (characterized by edema and erythema) through the stimulation of transient receptor potential cation channel subfamily V member 1 (TRPV1 receptors) on the sensory nerve endings in the skin. It is established that heat hyperalgesia (i.e., increased sensitivity to heat stimuli at the site of capsaicin application) results from peripheral sensitization, while mechanical hyperalgesia (i.e., increased sensitivity to mechanical stimuli outside the capsaicin area) is due to central sensitization.

Before capsaicin application, skin temperature is measured using an infrared thermometer. If the skin temperature is below 30°C, the area is covered with a blanket until the required skin temperature is reached. Capsaicin, 640 mg per cm² (corresponding to 5.76 mg of capsaicin in total), is transdermally applied to a 30 mm × 30 mm area on the volar side in the middle of both distal forearms of the participants. After 60 minutes, the capsaicin is removed, and the skin areas are treated with a cleansing gel. Spontaneous pain is then assessed using a Visual Analog Scale.

Subsequently spontaneous pain is determined using the Visual Analogue Scale. Since primary and secondary hyperalgesia is most pronounced at 1 hour after capsaicin application, the measurement of the allodynia distance, pinprick hyperalgesia, and the heat pain and perception thresholds are conducted in close temporal succession after 60 minutes.

After a 4-week wash-out phase, the third study visit is held. It included again the baseline measurement. Subsequently, the other substance is taken for 28 days. This is followed by the fourth study visit including the survey of the sensory parameters and the capsaicin pain model.

To investigate the influence of Boswellia serrata on the psyche, the participants answered four psychological questionnaires during all four study visits. These focused on depression, anxiety, sleep quality andwell-being. The names of the questionnaires are Becks-Depression-Index, Becks-Anxiety-Index, Pittsburgh Sleepquality-Index and WHO-5.

Sample size calculation:

As no previously published data are available as a source for an a priori calculation of the sample size, an estimate is made based on the following assumptions. The significance level is set at 0.05 and Beta at 0.2. For a two-sided paired t-test, a sample size of ten participants is sufficient to detect an effect size of ≥ 1. A dropout rate between 0.1 and 0.2 is anticipated, leading to a target sample size of n = 12 participants. Long-Illevich et al. used a similar study format with the same sample size planning in their publication.

Lang-Illievich K, Klivinyi C, Rumpold-Seitlinger G, Dorn C, Bornemann-Cimenti H. The Effect of Palmitoylethanolamide on Pain Intensity, Central and Peripheral Sensitization, and Pain Modulation in Healthy Volunteers-A Randomized, Double-Blinded, Placebo-Controlled Crossover Trial. Nutrients. 2022 Oct 1;14(19)

Statistics:

No data are available on the probability of a period effect. The probability of a carryover effect is low, as the washout interval of 28 days was chosen to be sufficiently long, as a HWZ of Boswellia serrata of approx. 2 h is assumed.

After completion of the data collection, descriptive statistics were performed (separately for treatment A and B as well as period 1 and 2). Continuous values were summarized using mean, median, standard deviation, minimum and maximum. The Shapiro-Wilk test is used to verify a possible normal distribution. This is followed by a comparison of the results of both periods and treatment series (AB vs. BA) as well as a check for a carryover effect (comparison of the first periods of treatments A and B using an unpaired t-test). The further statistical procedure depends, among other things, on the existence of a carryover effect and the completeness of the data. Accordingly, if the preconditions are met, either a linear mixed model (LMM; e.g. for missing values or dropouts) or an ANOVA (advantageous when considering period and subject effects) is used. If there is no normal distribution, a Wilcoxon signed rank test can be used. With a p-value <0.05, the null hypothesis was rejected. Qualitative data is evaluated using a chi-square test. The effect size is calculated by dividing the Z value by the square root of N.

Study substance:

The participants each receive 56 capsules containing either Boswellia serrata 300 mg (Wunschkapsel) or an optically identical placebo (veggie capsules, size 0, maltodextrin filler) manufactured in a pharmacy. It is taken at 24-hour intervals. The last dose is taken in the morning before the study visit. To increase adherence to therapy, an electronic reminder will be sent via cell phone. Capsules that have not been taken should be brought to the study visit after the respective intake interval.

Parameter:

Spontaneous pain:

Directly after the last heat application, the spontaneous pain is recorded using the VAS scale, which is used throughout the LKH Univ.-Klinikum Graz.

Allodynia:

Starting from the center of the thermal application, a von Frey filament (128 mN) is applied to the skin in 4 radial lines at a 5 mm interval, first from the inside to the outside, then from the outside to the inside, and the distance at which an unpleasant pointed sensation first occurs is determined. The 8 measurements are averaged.

Pinprick hyperalgesia:

By means of a pinprick with 256 mN a pointed stimulus is applied. The test site is 5 cm proximal to the center of the thermal stimulation area. A numerical scale (0-100) is used to measure how painful this stimulus is.

Heat pain and perception threshold:

The heat detection threshold and the heat pain threshold are determined according to the guidelines of the German Research Association for Neuropathic Pain, which involves heating the skin with TSA-II NeuroSensoryAnalyser. The test person can stop the heating by pressing a stop button. This should be done at the first time he/she notices that the skin is warming up (heat detection threshold) or at the time he/she notices a pulling, burning or pricking sensation in addition to the feeling of heat (heat pain threshold). The measurements are taken 3 times each and the results are averaged.

Conditioned pain modulation:

Conditioned pain modulation describes the function of the descending, pain-inhibiting system. First, the force with which pressure on the adductor pollicis brevis muscle of the non-dominant hand is not only perceived as pressure, but also as a stabbing, burning or pulling sensation is determined using a pressure gauge. Subsequently, the contralateral hand is immersed in ice water until the subject feels a pain intensity of NRS 40 (101-part scale). The pressure pain threshold is then immediately raised again.

Adverse effects:

Possible adverse effects are assessed and documented at each study visit. In addition, the subjects are informed about the necessity of immediate telephone contact in case of the occurrence of undesirable side effects.

Recruitment and informed consent:

Recruitment of participants is done by posting on notice boards at the ÖH an der Med-Uni Graz (main building) and the outpatient pain clinic

Participants are asked orally whether they participate in another study at the same time or whether a required period of time has elapsed since participation in another study. They confirm this with their signature.

A physician involved in the study will provide the information. Consent is then given by signing a written information sheet.

The investigation of pain and perception thresholds according to the specifications of the "German Research Association for Neuropathic Pain" is an established procedure in both human research and clinical investigation. No danger is to be expected for the individual test person.

The cutaneous capsaicin patch should only be applied to dry, intact (uninjured) skin and not on the face, over the hairline of the scalp, or near mucous membranes. Temporary local reactions at the application site, such as burning, mild pain (NRS 1-3), redness, and itching, are common or very common. Aside from acute local reactions at the application site, published non-clinical and clinical data on the 8% capsaicin patch do not show any specific safety concerns regarding skin exposure to capsaicin or its metabolites. If, contrary to expectations, participants experience severe pain (>NRS 6), the patch will be removed immediately, and the skin will be checked for signs of local burns. Participants who experience pain during or after the patch application will receive supportive treatment, such as local cooling (using a cold compress). The changes in pain sensitivity are strongly localized and normalize within a few hours.

If the individual test person is willing to be exposed to a pain stimulus for a limited period of time, there is no foreseeable risk for him/her.

Boswellia serrata marketed as a food supplement in accordance with EU Directive 2002/46/EC. In general, Boswellia serrata is considered a safe dietary supplement with no severe long-term side effects. Mild side effects such as diarrhea, abdominal pain, and vomiting may occasionally occur. However, there is no evidence of severe side effects associated with the use of Boswellia serrata.

List of side effects according to their frequency (from most common to rare): Abdominal pain, Diarrhea, Loss of appetite, Heartburn, Nausea/vomiting, Allergic reaction to boswellic acid.

Contraindications include known allergies of boswellia acids. Due to a lack of studies, it is not recommended for use during pregnancy and breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years

Exclusion Criteria:

* Not pregnant or breastfeeding
* No renal or liver insufficiency
* No neurological/dermatological/cardiovascular diseases
* No chronic pain and/or use of analgesics
* No use of anticoagulants
* No use of antidepressants
* No use of MAO inhibitors
* No use of St. John's Wort
* No use of medications affecting the CYP mechanism
* No allergies to Boswellia serrata or capsaicin"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in spontaneous pain intensity | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  is measured on a visual analogue scale (0 means no pain and 10 means the worst imaginable pain)

SECONDARY OUTCOMES:
Change in Allodynia | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  Starting from the center of the capsaicin application, a von Frey filament (128 mN) is applied to the skin in four radial lines at 5 mm intervals, first from the outside to the inside, followed by a measurement from the inside to the outside. The distance at which a sharp unpleasant sensation first occurre or cease is determined. The eight measurements are averaged. A low score means a worse outcome, a higher score a better outcome.
Change in Hyperalgesia | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  When testing temporal summation, the perceived pain intensity of a single pinprick stimulus iscompared to a sequence of 10 pinprick stimuli of the same force repeated at a rate of 1/s (256 mN). A train of pinprick stimuli will be given within a small area of 1 cm² approximately 5 cm proximal to the middle of the capsaicin stimulation area. The subject will be asked to give a pain rating representing the pain at the end of the train using a numerical rating scale (0-100). The wind-up ratio (WUR) will be calculated as the mean pain rating of three trains divided by the mean pain rating for the single stimuli. A low score means good outcome, a higher score a worse outcome (0-100).
Change in heat detection threshold | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  The skin will be heated with a TSA-II Neuro Sensory Analyzer (Medoc Ltd. Advanced Medical Systems, Ramat Yishai, Israel). The proband is instructed to stop the heating via a stop button once he noticed the increase in temperature (heat detection threshold). Each measurement will be performed three times, and the results will be averaged. Measured in degrees C° A low score means worse outcome, a higher score a good outcome.
Change in heat pain threshold | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  measured in degrees C°
Change in conditioned pain modulation | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  measures the descending analgesic System with the help of a pressure algometer in kg
Change of depression score | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  Change of questionnaire BDI-II score. A BDI-II score is classified by total score ranges: 0-13 (Minimal), 14-19 (Mild), 20-28 (Moderate), and 29-63 (Severe), with higher scores indicating greater severity of depressive symptoms. Each of the 21 items on the self-report questionnaire is scored from 0 to 3, and the total score is the sum of all 21 items.
Change of anxiety score | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  Change of questionnaire BAI score. The Beck Anxiety Inventory (BAI) score ranges from 0 to 63 and shows how severe a person's anxiety symptoms are. Each question is scored with 0-3 points. Higher scores mean more severe anxiety.
  0-7 = Minimal anxiety 8-15 = Mild anxiety 16-25 = Moderate anxiety 26-63 = Severe anxiety
Change of sleep quality score | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  The Pittsburgh Sleep Quality Index (PSQI) measures the quality of a person's sleep over the past month. The total PSQI score ranges from 0 to 21. Higher scores mean worse sleep quality.
  0-5 = Good sleep quality 6-10 = Moderate sleep difficulties 11-21 = Poor sleep quality / severe difficulties
Change of well-being score | Day 0 -->Day 28 before capsaicin pain model --> Day 28 1 hour after capsaicin pain model --> Day 56 -->Day 84 before capsaicin pain model -->Day 84 1 hour after capsaicin pain model
  The WHO-5 Well-Being Index measures emotional well-being over the past two weeks. It has 5 questions, each scored from 0 (at no time) to 5 (all of the time). The total raw score ranges from 0 to 25, then it's multiplied by 4 to give a final score out of 100. A low score means worse outcome, a higher score better outcome.
  0-50 = Poor well-being 51-100 = Good well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No